CLINICAL TRIAL: NCT06018363
Title: Allogeneic B7-H3 CAR-γδT Cell Therapy Recurrent/Progressive High Grade Glioma（R/R HGG）
Brief Title: Clinical Study on the Treatment of Malignant Brain Glioma by QH104 Cell Injection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dushu Lake Hospital Affiliated to Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QH10401-GC-01（0）
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Brain Gliomas; High-Grade Gliomas; GBM
Keywords: B7-H3; CAR-γδT; allogeneic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with R/R HGG (Experimental)
  Interventions: Biological: Allogenic B7-H3 CAR-γδT cell(QH104)

INTERVENTIONS:
Biological: Allogenic B7-H3 CAR-γδT cell(QH104) — Dose escalation (3+3) : dose 1 (1 × 10^7 CAR+cells) , dose 2 (3 × 10^7 CAR+cells), dose 3 (6× 10^7 CAR+cells), once every 4 weeks via an Ommaya reservoir or intrathecal administration.
  Dose expansion 1: dose of RP2D, once every 4 weeks via an Ommaya reservoir or intrathecal administration.
  Dose expansion 2: 3 × 10^7 CAR+cells, every two weeks for three consecutive months, then changed to once every 4 weeks via an Ommaya reservoir or intrathecal administration.

SUMMARY:
B7-H3 is expressed at low levels in normal tissues but overexpressed in various tumor tissues. The ubiquitous expression of B7-H3 in tumors of different grades is a key feature for brain gliomas. The immunohistochemistry study showed that B7-H3 is abundantly expressed on both glioma (especially high-grade glioma) cells and tumor-associated endothelial cells. For GBM, the expression of B7-H3 is intensely positive, especially on tumor cells and vascular endothelial cells, which makes B7-H3 a potential immunotherapeutic target.

γδ T cells recognize tumor cells without being restricted by MHC molecules, and thus can be used in allogeneic therapy without the risk of causing graft-versus-host disease.

This study is an open-label, single-arm, dose-escalation and dose-expansion clinical study aimed at evaluating the safety and efficacy of allogeneic B7-H3 CAR γδT in patients with malignant glioma.

ELIGIBILITY:
Inclusion Criteria:

* 1)Age 18-70 years old (both ends included), both male and female;
* 2)At least one evaluable lesion, with previous biopsy or histopathological confirmation of high-grade glioma (WHO grade 3-4), and after comprehensive treatment, imaging examination indicates continued progression or recurrence;
* 3) The pathological tissues removed by surgery can be used for immunohistochemical detection of target proteins (paraffin sections should be within half a year), and the expression of B7-H3 is positive;
* 4) KPS ≥ 60 points;
* 5)Expected survival > 3 months;
* 6)Substantially normal bone marrow reserve function and normal liver and renal function (laboratory tests need to be fulfilled before receiving QH104 Cell Injection for the first time):White blood cell count (WBC) ≥ 3 x 10^9/L;Lymphocyte count (LY) ≥ 0.8 x 10^9/L;Hemoglobin (Hb) ≥ 90g/L;Platelet (PLT) ≥80×10^9/L;Albumin transaminase (ALT) & albumin transaminase (AST) <1.5×ULN;Serum creatinine (Cr) <1.5 x ULN;Total bilirubin < 1.5 x ULN;PT & PTT ≤ 1.25 x ULN.
* 7)No obvious hereditary diseases;
* 8)Normal cardiac function with cardiac ejection index >55%;
* 9)No bleeding and coagulation disorders;
* 10)Women of childbearing age (15-49 years old) must have had a pregnancy test with a negative result within 7 days prior to the start of treatment, and subjects are willing to use contraception during the clinical trial and for 3 months after the last cell infusion;
* 11) Sign the informed consent form.

Exclusion Criteria:

* 1)Pregnant and lactating women;
* 2)Those with organ failure:Heart: Class III and IV;Liver: up to grade C of the Child-Turcotte Liver -Function Classification;Kidney: chronic kidney disease stage 4 or above; renal insufficiency stage III or above;Lungs: symptoms of severe respiratory failure with involvement of other organs;Brain: central nervous system abnormalities or impaired consciousness;
* 3)patients with combined second tumors;
* 4)patients with active hepatitis B or C virus, HIV infection, or other untreated active infection;
* 5)any severe, uncontrolled systemic autoimmune disease or any unstable systemic disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis, Crohn's disease, and temporal arteritis;
* 6)Current systemic use of steroid cell (except for recent or current use of inhaled steroids) substances;
* 7) have a chronic disease requiring immunologic or hormonal therapy;
* 8) have an allergy to immunotherapy and related cells;
* 9) 10)Patients with a history of organ transplantation or who are awaiting organ transplantation;
* 10)Participation in other clinical trials within the previous 30 days;
* 11)Those who are not suitable for clinical trials for other reasons in the opinion of the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | 12 months
  AE is defined as any adverse medical event from the date of the cell infusion to 12 months after B7-H3 CAR-γδT cells infusion. Among them, cytokine release syndrome (CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria, graft-versus-host disease (GVHD) according to criteria defined by the Mount Sinai Acute GVHD International Consortium. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1:Incidence of Dose-Limiting Toxicities (DLTs) | 28 days after the first dose of B7-H3 CAR-γδT cells
  DLT was defined as B7-H3 CAR-γδT cells-related events with onset within first 28 days following infusion
Phase 1:Maximum tolerated dose (MTD) | 28 days after the first dose of B7-H3 CAR-γδT cells
Phase 1: Recommended phase 2 dose (RP2D) | 28 days after the first dose of B7-H3 CAR-γδT cells

SECONDARY OUTCOMES:
Pharmacokinetics: copy number of B7-H3 CAR-γδT cells in cerebrospinal fluid(CSF) | 28 days after the first dose of B7-H3 CAR-γδT cells
Pharmacodynamics: Peak level of cytokines in CSF | 28 days after the first dose of B7-H3 CAR-γδT cells
Phase 2: Overall survival (OS) | 6 months, 9 months and 12 months
Phase 2: Progression Free Survival (PFS) | 6 months
Disease Control Rate (DCR) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dushu Lake Hospital Affiliated to Soochow University, Suzhou, Jiangsu, China